CLINICAL TRIAL: NCT01339117
Title: Delivered Dietary Intervention for Children With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: NASPGHAN Foundation (Other Government)
Responsible Party: Principal Investigator, Bruno Chumpitazi, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-28050
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain
Keywords: irritable bowel syndrome; children; chronic abdominal pain; recurrent abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fermentable substrate diet (Experimental): High fermentable substrate diet provided for two days
  Interventions: Other: High fermentable substrate diet
- Low fermentable substrate diet (Experimental): Low fermentable substrate diet provided for two days
  Interventions: Other: Low fermentable substrate diet

INTERVENTIONS:
Other: Low fermentable substrate diet — Diet low in fermentable oligosaccharides, disaccharides, monosaccharides, and polyols.
  Arms: Low fermentable substrate diet
Other: High fermentable substrate diet — Diet high in fermentable oligosaccharides, disaccharides, monosaccharides and polyols
  Arms: High fermentable substrate diet

SUMMARY:
The purpose of this study is to determine whether a specific diet may help children with irritable bowel syndrome.

DETAILED DESCRIPTION:
Many children experience stomach pain or discomfort at some point during their lives. Some children have belly discomfort frequently while others rarely have this problem. There have been very few studies to test treatments for recurrent stomach discomfort in children. Recently, studies in adults with recurrent stomach discomfort suggest that diet changes may help. Currently, we do not know if these same diets will work in children with the same problem.

In this study, two different diets will be provided (delivered) for two days with at least 5 days in between each provided diet. The child's symptoms will be recorded over the two days of each diet. Children will be asked to capture samples of their breath during the last day of the each two day delivered diet. Stool samples will also be collected.

ELIGIBILITY:
Inclusion Criteria:

Must include all of the following:

1. Children between the ages of 7-17 years;
2. Meet the criteria for IBS based on the Questionnaire on Pediatric Gastrointestinal Symptoms Rome III Version, including pain/discomfort a minimum of twice per week;
3. Negative physician evaluation for an organic etiology of the pain within the past year

Exclusion Criteria:

Will include any of the following:

1. Diabetes or other disease process requiring specialized dietary management;
2. Malnutrition or obesity (BMI >95%);
3. Inability to eat by mouth;
4. Antibiotic or medicinal probiotic usage within the past 3 months (excluding yogurt);
5. Neuromodulator (e.g. amitriptyline) usage within the past 3 months
6. Start of, or change in gastrointestinal medication (e.g. laxative) dose that may cause or ameliorate abdominal symptoms within the past month

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Average daily abdominal pain frequency | 9 days (2 dietary intervention periods)
  Comparisons of abdominal pain frequency (number of abdominal pain episodes per day) will be made between each two day dietary period spanning a 9 days.

SECONDARY OUTCOMES:
Abdominal pain severity | 9 days (2 dietary intervention periods)
  The severity of abdominal pain episodes will be measured on a 1-10 (10 being most severe) ordinal scale. Average severity per abdominal pain episode during each two day dietary period will be compared over 9 days.
Hydrogen gas production | 9 days (2 dietary intervention periods)
  Daily hydrogen gas production (parts per million) will be compared between each 2 day dietary intervention period over 9 days.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno P Chumpitazi, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Children's Nutrition Research Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Chumpitazi BP, Cope JL, Hollister EB, Tsai CM, McMeans AR, Luna RA, Versalovic J, Shulman RJ. Randomised clinical trial: gut microbiome biomarkers are associated with clinical response to a low FODMAP diet in children with the irritable bowel syndrome. Aliment Pharmacol Ther. 2015 Aug;42(4):418-27. doi: 10.1111/apt.13286. Epub 2015 Jun 24. PMID 26104013